CLINICAL TRIAL: NCT07024485
Title: Effect of Augmented Reality Animations in Nursing Smoking Cessation Training for Nursing Students: A Randomized Controlled Trial
Brief Title: Augmented Reality Animations for Smoking Cessation Counseling Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EA250324
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation Counseling Ability and Practice
Keywords: AR animation; nursing students; smoking cessation training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinding technique will be used to conceal the allocation. Participants will not know which group they are in as placebo messages will be introduced. Using a central allocation web-based-controlled randomization, outcome assessors and data analysts will be blind to group allocation, only the principal investigator will be aware of who belongs to the control and intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Teaching format: Tutorial includes Augmented Reality (AR) animations Learning materials: Watch 4 smokers' real-life scenario videos + read case texts + interact with AR animations Discussion preparation: Develop quit plan using 5As model and AR animations; prepare for role-play Role-play and simulation: Use AR visuals to support counseling demonstration; each group role-plays using 5As model Technology/tools required:Smartphone with browser (iOS/Android); no app download needed
  Interventions: Device: AR animations and 5As model based on smoking cessation counseling Knowledge-Attitude-Practice (KAP)
- Control group (Placebo Comparator): Teaching format: Traditional tutorial without AR animations Learning materials: Watch 4 smokers' real-life scenario videos + read case texts only Discussion preparation: Develop quit plan using 5As model; prepare for role-play (no AR used) Role-play and simulation: Role-play based on text and video only; 5As model used Technology/tools required:No specific technology required
  Interventions: Device: 5As model based on smoking cessation counseling Knowledge-Attitude-Practice (KAP)

INTERVENTIONS:
Device: AR animations and 5As model based on smoking cessation counseling Knowledge-Attitude-Practice (KAP) — The intervention group received a tutorial that incorporated Augmented Reality (AR) animations alongside conventional teaching materials. In addition to watching four real-life smoker scenario videos and reading corresponding case texts, students used their smartphones to interact with AR animations that visualized the physiological effects of smoking (e.g., lung cancer, vascular disease, aging). These animations were used during group discussions and role-play sessions, helping students to assess smokers' knowledge, illustrate health risks, and tailor counseling plans using the 5As model. The AR experience was designed to enhance learning engagement, emotional connection, and self-efficacy in delivering smoking cessation counseling.
  Arms: Intervention group
Device: 5As model based on smoking cessation counseling Knowledge-Attitude-Practice (KAP) — The control group, received a conventional tutorial without the use of AR technology. They watched the same four smoker scenario videos and read the same case texts, then engaged in small group discussions and role-play activities to develop quit plans using the 5As counseling model. However, unlike the intervention group, their learning process relied solely on textual and video materials, without the immersive or interactive elements provided by AR. This approach represents standard smoking cessation training methods commonly used in nursing education.
  Arms: Control group

SUMMARY:
This proposed study aims to develop augmented reality (AR) based intervention during the smoking cessation counselling(SCC) training for master nursing students in the University of Hong Kong.

Hypotheses to be tested: (1) AR animations can improve nursing students' knowledge, skills in SCC compared to conventional teaching methods. (2)Student satisfaction and engagement with AR-based learning can be improved. (3) The training will increase master nursing students' self-efficacy to application of 5As SCC skill.

The study is a pragmatic randomized controlled trial (RCT) with a 1:1 allocation ratio, using AR animations for intervention and control groups. The intervention group receives messages related to SCC, while the control group receives generic mental health information. The subjects are MN students enrolled in the "Tobacco Dependency Nursing Intervention and Management" course.

The study uses various tools for measurement, including Providers Smoking Cessation Training Evaluation(ProSCiTE), and The Instructional Materials Motivation Survey (IMMS). The main outcome measures include SCC practice frequency,SCC knowledge score, SCC attitude score, and SCC practice score.

Data will be entered into SPSS for Windows (version 20) for analysis. Descriptive statistics including frequency, percentage, and mean will be used to summarize the outcomes and other variables. By intention-to-treat analysis, participants who are lost or refuse the follow-up will be treated as no change in the training outcomes. Chi-square tests and t-tests will be used to compare outcomes between intervention and control groups. The effect size, Cohen's d, will be computed for the standardized mean of the pre-post differences, both with and without adjustment for baseline characteristics. Additionally, Cohen's f will be calculated to assess the magnitude of the intervention effect in the linear mixed models. These models, which account for multiple observations per subject and clustering effects, will be used to analyze the intervention's impact on self-efficacy, motivation, and KAP. Both the main effect (group allocation) and interaction effect (group × time) will be examined to determine the intervention's effectiveness.

DETAILED DESCRIPTION:
This study proposes the development and evaluation of an augmented reality (AR)-based intervention integrated into the smoking cessation counselling (SCC) training for Master of Nursing (MN) students at the University of Hong Kong. The goal is to enhance students' competencies in applying the 5As framework (Ask, Advise, Assess, Assist, Arrange) in tobacco dependency interventions.

This study adopts a two-arm, waitlist-controlled, pragmatic randomized controlled trial (RCT) design with a 1:1 allocation ratio. Eligible participants are MN students enrolled in the "Tobacco Dependency Nursing Intervention and Management" course (NURS8205) in the Spring 2025 semester. Participants will be randomly assigned into intervention and control groups, stratified by tutorial group, and balanced across four trained facilitators.

Intervention Group: Receives the AR-enhanced SCC tutorial, which includes the following components:

1. Viewing videos of four simulated smoker-patient scenarios.
2. Reviewing case-based written materials.
3. Interacting with AR animations embedded in the learning platform, which visualize behavioral counselling techniques and simulate patient-provider communication aligned with the 5As model.

Control Group: Receives the standard tutorial format, which includes:

1. Viewing the same four smoker videos.
2. Reading the same case-based written materials.
3. No AR content is provided; instead, supplementary materials unrelated to SCC will be included to maintain time-equivalent exposure.

The intervention has been developed to align with adult learning theory and aims to enhance knowledge retention, skill application, and learner engagement. Tutors leading both intervention and control sessions will receive standardized training to ensure consistency.

Measurement and Data Collection Assessments will be conducted at baseline (pre-intervention), immediately post-intervention, and follow-up at 2-month post-intervention.

Key instruments include:

1. Providers Smoking Cessation Training Evaluation (ProSCiTE): This validated tool will be used to assess four constructs: knowledge, attitude, self-efficacy, and SCC behavior. It serves as the primary tool for evaluating changes in KAP and self-efficacy.
2. Instructional Materials Motivation Survey (IMMS): Based on Keller's ARCS model (Attention, Relevance, Confidence, Satisfaction), IMMS will measure students' engagement, satisfaction, and motivation related to the learning materials.

Data Analysis Data will be analyzed using SPSS for Windows version 20. Descriptive statistics (means, SDs, frequencies, and percentages) will summarize baseline characteristics and outcome variables.

Intention-to-treat analysis will be applied, where participants lost to follow-up will be assumed to have no change from baseline scores.

Independent t-tests and chi-square tests will compare primary and secondary outcomes between groups.

Effect sizes will be calculated:

Cohen's d for standardized pre-post mean differences. Cohen's f for evaluating the intervention effect size in linear mixed-effects models, which will control for repeated measures and potential clustering effects (e.g., by tutorial group or tutor).

These models will assess both:

Main effect of the intervention (between-group differences). Interaction effect between group and time (i.e., whether change over time differs between groups).

Expected Impact

It is anticipated that the AR-based intervention will lead to:

Increased self-efficacy in delivering SCC using the 5As model. Enhanced knowledge and positive attitudes toward smoking cessation. Improved SCC practice behaviors during clinical placements. Greater learner motivation and satisfaction compared to traditional tutorial methods.

This innovative pedagogical approach aligns with contemporary nursing education trends and aims to equip future nurses with effective behavioral counselling skills to address tobacco dependence.

ELIGIBILITY:
Inclusion Criteria:

* master nursing students (1-2 years)
* able to read, understand, and write in English
* willing to participate in this study

Exclusion Criteria:

- students who have taken any training courses in the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | T0: Baseline (Day 1 of course) T1: Pre-tutorial (Immediately before the tutorial session) T2: Post-tutorial (Immediately after the tutorial session) T3: Follow-up (2 months after the tutorial session)
  Self-efficacy in applying the 5As framework of SCC will be measured using the Providers Smoking Cessation Training Evaluation (ProSCiTE) scale. This validated tool includes subscales measuring knowledge, attitude, self-efficacy, and behavior. The self-efficacy subscale evaluates the confidence of nursing students in delivering SCC.
  Scoring:
  Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  Minimum score: 13 Maximum score: 65 Higher scores indicate greater self-efficacy in providing SCC.

SECONDARY OUTCOMES:
Learning motivation and satisfaction | T0: Baseline (Day 1 of the course) T1: Pre-tutorial (Immediately before the tutorial session) T2: Post-tutorial (Immediately after the tutorial session) T3: Follow-up (2 months after the tutorial session)
  Learning motivation and satisfaction will be assessed using the Instructional Materials Motivation Survey (IMMS). This validated instrument consists of 36 items designed to measure learners' reactions to instructional materials, based on Keller's ARCS model of motivation (Attention, Relevance, Confidence, and Satisfaction).
  Subscales:
  Attention (12 items) Relevance (9 items) Confidence (9 items) Satisfaction (6 items)
  Scoring:
  Each item is rated on a 5-point Likert scale from 1 (not true) to 5 (very true). Negatively worded items are reverse-scored.
  Minimum total score: 36 Maximum total score: 180 Higher scores indicate greater motivation and satisfaction with the learning experience.
knowledge, attitude, and behavior in Smoking Cessation Counselling | T0: Baseline (Day 1 of the course) T1: Pre-tutorial (Immediately before the tutorial session) T2: Post-tutorial (Immediately after the tutorial session) T3: Follow-up (2 months after the tutorial session)
  Knowledge, attitude, and behavior (KAB) related to smoking cessation counselling (SCC) will be assessed using the Providers Smoking Cessation Training Evaluation (ProSCiTE) scale. This validated instrument is designed to evaluate the effectiveness of SCC training among healthcare providers. In this study, the subscales measuring knowledge, attitude, and behavior will be used to assess master nursing students' understanding, perceptions, and application of the 5As framework in SCC.
  Scoring:
  Knowledge subscale:
  Minimum score: 0 Maximum score: 14 Higher scores indicate greater factual knowledge.
  Attitude and Behavior subscales:
  Minimum score: 8 ,19 Maximum score: 40, 95 Higher scores indicate more positive attitudes and greater engagement in SCC-related behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong KongLKS Faculty of MedicineHong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 5 years.
Access Criteria: Research data and documentation will be available upon request.